CLINICAL TRIAL: NCT04422171
Title: A 12-month Real Life Study of IBD Patients Under Stable Steroid Free Clinical and Biological Remission Switched From Adalimumab Originator Humira® to One of Its Biosimilar: Amgevita®,Hulio®,Hyrimoz® or Imraldi®.
Brief Title: A 12-month Real Life Study of IBD Patients Switched From Adalimumab Originator Humira® to One of Its Biosimilar
Acronym: Rhoneswitch
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC19.379; 2020-A00494-35 (Other: ID RCB)
Record Dates: First submitted 2020-06-04; First posted 2020-06-09 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: IBD Patients, Originator Treatment, Biosimilar, Switch Back

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Biosimilars represent great potential in cost saving and reinvestment opportunities in healthcare. Biosimilars of adalimumab appear to be clinically equivalent to the reference product in patients with rheumatoid arthritis and psoriasis. No data are currently available in IBD patients. Real-life data are needed.

Minimizing the switch back is another clinical challenge in the current area of biosimilars. The primary objective of Rhoneswitch is to describe the magnitude of patient's switch back defined as a deterioration of symptoms without objective identification of disease activity, 12 months after the switch from ada originator Humira®.

The primary endpoint is to assess the percentage of patients who switch back to originator therapy Humira® 12 months after switching from ada Humira® to ada Bs: Amgevita® ,Hulio®, Hyrimoz® or Imraldi® in IBD patients without any objective markers of inflammation.

DETAILED DESCRIPTION:
The subject will be include during usual hospital consultation after reviewing inclusion/exclusion criteria and obtain non opposition. Data will be collected during 3 usual hospital consultations: at month 3, month 6, and month 12. The end of study will be at month 12 or at premature termination.

Questionnaires will be done in addition during all usual hospital consultations.

ELIGIBILITY:
INCLUSION CRITERIA

* Documented diagnosis of CD or UC established on the basis of standard clinical, endoscopic and histological criteria at least 3 months prior to inclusion.
* Inactive CD or UC outpatients are defined per clinical assessment as an Harvey Bradshaw Index (HBI) score ≤4 for CD patients and a Partial Mayo Score (PMS) ≤2 with each sub-score of 1 or less for UC and/or according to ECCO classification (Sturm 2019) within previous 3 months, demonstrating an adequate clinical remission to ada originator
* May be receiving the following drugs (but must remain on stable dose for 10 weeks):

  * Oral 5-aminosalicylates (ASA) compounds or rectal formulations of 5ASA provided the dose to be stable at least 4 weeks before switching
  * Azathioprine, 6-MP or methotrexate provided the dose has been stable for 4 weeks prior to inclusion (dose must remain stable for 10 weeks after switching)
* Non opposition required

EXCLUSION CRITERIA

* Diagnosis of indeterminate colitis, ischaemic colitis, fulminant colitis
* Current use of another TNF inhibitor included (but not limited to) infliximab, certolizumab, golimumab
* Current use of vedolizumab or ustekinumab
* Current use of JAK inhibitors or S1P modulators
* Current use of oral corticosteroids
* Active flaring CD or UC patients defined as a HBI > 4 for CD and a PMS>1 for UC and/or concomitant CS medication
* Pregnancy or breast feeding
* Subject under guardianship or subject deprived of liberty

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: IBD Patients (Ulcerative Colitis and Crohn's disease) under stable (more than 3 months) steroid free clinical and biological remission with adalimumab.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-06-19 (Actual); Primary Completion 2021-06-18 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
Magnitude of patient's switch back defined as a deterioration of symptoms without objective identification of disease activity, 12 months after the switch from ada originator Humira®. | 12 months
  Percentage of patients who switch back to originator therapy Humira® 12 months after switching from ada Humira® to ada Bs: Amgevita® ,Hulio®, Hyrimoz® or Imraldi® in IBD patients without any objective markers of inflammation.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Mathieu, Principal Investigator — CHU Grenoble Alpes
Locations (1):
- Chu Grenoble Alpes, Grenoble, France